CLINICAL TRIAL: NCT01123460
Title: Measurement of Potential Biomarkers Predicting Erlotinib Response
Brief Title: Biomarkers Predicting Response in Patients With Non-Small Cell Lung Cancer Previously Treated With Erlotinib Hydrochloride
Status: Completed | Type: Observational
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Other Study IDs: CDR0000670992; ECOG-E3503T2
Record Dates: First submitted 2010-05-13; First posted 2010-05-14 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Lung Cancer
Keywords: non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Enzyme-Linked Immunosorbent Assay

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Other: enzyme-linked immunosorbent assay
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood in the laboratory from patients receiving erlotinib hydrochloride may help doctors learn more about the effects of erlotinib hydrochloride on cells. It may also help doctors understand how well patients respond to treatment.

PURPOSE: This research study is studying biomarkers predicting response in patients with non-small cell lung cancer previously treated with erlotinib hydrochloride.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate whether serum NGAL, MMP-9, NGAL/MMP-9 complex, and soluble E-cadherin can be utilized as biomarkers to predict response in patients with non-small cell lung cancer treated with erlotinib hydrochloride.

OUTLINE: Serum samples are analyzed for NGAL, MMP-9, NGAL/MMP-9, and soluble E-cadherin by ELISA and Luminex assays.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of non-small cell lung cancer
* Received erlotinib hydrochloride on clinical trial ECOG-E3503

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples submitted for research from patients enrolled on E3503
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2010-04-12 (Actual); Primary Completion 2010-06-12 (Actual); Study Completion 2010-06-12 (Actual)

PRIMARY OUTCOMES:
Baseline serum NGAL, MMP-9, NGAL/MMP-9 complex, and soluble E-cadherin levels as predictors of erlotinib hydrochloride response | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Steven M. Dubinett, MD, Principal Investigator — Jonsson Comprehensive Cancer Center